CLINICAL TRIAL: NCT02124044
Title: Safety, Tolerability, and Efficacy of Daclatasvir and Asunaprevir, With or Without BMS-791325, in Subjects Coinfected With HIV-HCV
Brief Title: Safety, Tolerability, and Efficacy of Asunaprevir and Daclatasvir in Subjects Coinfected With HIV-HCV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 140065; 14-CC-0065 (Other: National Institutes of Health)
Record Dates: First submitted 2014-04-25; First posted 2014-04-28 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2017-05-16 (Actual); Status verified 2017-04

CONDITIONS: HIV-HCV
Keywords: Coinfection; HCV Genotype 1b; Interferon Free therapy; Liver Biopsy; Virological Response
MeSH Terms: conditions — Coinfection | interventions — asunaprevir; daclatasvir; 8-cyclohexyl-N-((dimethylamino)sulfonyl)-1,1a,2,12b-tetrahydro-11-methoxy-1a-((3-methyl-3,8-diazabicyclo(3.2.1)oct-8-yl)carbonyl)cycloprop(d)indolo(2,1-a)(2)benzazepine-5-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HIV/HCV GT-1b, 24 wks ASV/DCV (Experimental): Oral treatment with Asunaprevir 100mg (ASV), twice daily, and Daclatasvir 60mg (DCV), once daily, for 24 weeks in HIV/HCV genotype 1b patients
  Interventions: Drug: Asunaprevir and Daclatasvir
- HIV/HCV GT-1a/1b, 12 wks ASV/DCV with BMS-791325 (Experimental): Oral treatment with Asunaprevir 200mg (ASV), Daclatasvir 30 mg (DCV) and BMS-791325 75 mg in a fixed dose combination pill (FDC), twice daily, for 12 weeks in HIV/HCV genotype 1a or 1b patients
  Interventions: Drug: Asunaprevir and Daclatasvir with BMS-791325

INTERVENTIONS:
Drug: Asunaprevir and Daclatasvir — Oral treatment with Asunaprevir 100mg (ASV), twice daily, and Daclatasvir 60mg (DCV), once daily, for 24 weeks in HIV/HCV genotype 1b patients
  Other Names: Asunaprevir (ASV) and Daclatasvir (DCV)
  Arms: HIV/HCV GT-1b, 24 wks ASV/DCV
Drug: Asunaprevir and Daclatasvir with BMS-791325 — Oral treatment with Asunaprevir 200mg (ASV), Daclatasvir 30 mg (DCV) and BMS-791325 75 mg in a fixed dose combination pill (FDC), twice daily, for 12 weeks in HIV/HCV genotype 1a or 1b patients
  Other Names: Asunaprevir (ASV) and Daclatasvir (DCV) and BMS-791325 (Beclabuvir)
  Arms: HIV/HCV GT-1a/1b, 12 wks ASV/DCV with BMS-791325

SUMMARY:
Chronic hepatitis C virus (HCV) infection is a major public health problem with an estimated 180 million people infected worldwide. In the United States an estimated 4.1 million people are infected and HCV is the principal cause of death from liver disease and leading indication for liver transplantation. Within HIV/HCV co-infected patients, liver disease due to Hepatitis C progresses even more rapidly. While combination of ribavirin (RBV) and pegylated interferon (PEG) in combination with boceprevir/telaprevir is the currently recommended therapy for chronic HCV infection and has superior cure rates compared to PEG+RBV alone in HCV monoinfected patients, treatment is still associated with a high incidence of adverse events (AEs), discontinuations and poor cure rates in several populations. Within the HIV/HCV co-infected population treatment for HCV remains complicated given drug interactions between anti-retrovirals and HCV protease inhibitors, in addition to the extensive side-effects due to PEG +RBV alone. Recent studies have demonstrated that the use of a combination of anti-virals which target HCV without interferon (IFN) can cure HCV, without additional toxicities. These novel therapies that do not rely on an IFN backbone may additionally enhance cure rates in HIV/HCV co-infected, a population which has historically been difficult to cure.

The findings from this study will aid in the understanding of antiviral and host responses and determinants of response to an IFN free regimen in HIV/HCV co-infected patients.

DETAILED DESCRIPTION:
Chronic hepatitis C virus (HCV) infection is a major public health problem with an estimated 180 million people infected worldwide. In the United States an estimated 4.1 million people are infected and HCV is the principal cause of death from liver disease and leading indication for liver transplantation. Within HIV/HCV co-infected patients, liver disease due to Hepatitis C progresses even more rapidly. While combination of ribavirin (RBV) and pegylated interferon (PEG) in combination with boceprevir/telaprevir is the currently recommended therapy for chronic HCV infection and has superior cure rates compared to PEG+RBV alone in HCV monoinfected patients, treatment is still associated with a high incidence of adverse events (AEs), discontinuations and poor cure rates in several populations. Within the HIV/HCV co-infected population treatment for HCV remains complicated given drug interactions between anti-retrovirals and HCV protease inhibitors, in addition to the extensive side-effects due to PEG +RBV alone. Recent studies have demonstrated that the use of a combination of anti-virals which target HCV without interferon (IFN) can cure HCV, without additional toxicities. These novel therapies that do not rely on an IFN backbone may additionally enhance cure rates in HIV/HCV co-infected, a population which has historically been difficult to cure.

This is an open label study to assess the safety, tolerability and efficacy of two regimens for the treatment of HCV, asunaprevir (ASV) 100 mg BID and daclatasvir (DCV) 60 mg daily (selective HCV NS3 and NS5A inhibitors respectively) in 10 HIV/HCV genotype 1b co-infected treatment-naive and treatment experienced individuals and DCV + ASV + BMS-791325 administered as a fixed dose combination (FDC) pill in 20 HIV/HCV GT 1a or 1b coinfected treatment-naive and treatment experienced individuals.

The findings from this study will aid in the understanding of antiviral and host responses and determinants of response to an IFN free regimen in HIV/HCV co-infected patients.

ELIGIBILITY:
* INCLUSION CRITERIA

Subjects who meet the following criteria are eligible to enter the study:

1. Eighteen years of age or older at screening
2. Naive to treatment for hepatitis C or treatment experienced on previous IFN-containing treatment for chronic HCV infection. Patients who have been re-infected with HCV are excluded.
3. Women are allowed to participate if they agree to always use at least two forms of birth control. One form must be barrier protection (i.e., condom or female condom) and the other is to meet one of the criteria below:

   1. Non-childbearing potential status (i.e., physiologically incapable of becoming pregnant)

      - Has had a hysterectomy or

      - Has had a bilateral oophorectomy or

      - Is post-menopausal (age greater than or equal to 50 and a demonstration of a total cessation of menses for greater than or equal to 1 year) or

      - Has had a bilateral tubal ligation or fallopian tube inserts
   2. Childbearing potential status women must have a negative serum pregnancy test at screening and agree to use an acceptable form of birth control, such as any of the following:

      - Complete abstinence from sexual intercourse 2 weeks prior to administration of the study drug until completion of the follow-up procedures and at least 5 weeks (women) after the last dose of the study drugs.

      - Vasectomized partner in reliably monogamous relationship.
      * An intrauterine device (IUD) 2 weeks prior to administration of the study drugs continuously until completion of the follow-up procedures and at least 5 weeks after the last dose of the study drugs.
      * Double contraceptive method (condom or occlusive cap [diaphragm or cervical/vault caps]; spermicidal foam/gel/film/cream/suppository).
      * Oral, implantable, transdermal, or injectable or any other form of hormonal contraceptives are NOT an acceptable form of contraception for females on this study.
4. Men are allowed to participate if they agree to use at least 2 forms of birth control. One form must be barrier protection (i.e., condom or female condom) and the other is to meet one of the criteria below:

   1. Are sterile or
   2. Agree to use at least one of the following approved methods of contraception 2 weeks prior to administration of the study drug until the completion of the followup procedures and at least 14 weeks after the last dose of the study drugs:

      * A male condom with spermicide.
      * A sterile sexual partner.
      * A female sexual partner who has an IUD.
      * A female sexual partner using a female condom with spermicide, intravaginal system (e.g., NuvaRing[registered]), diaphragm with spermicide, cervical cap with spermicide, or oral, implantable, transdermal, or injectable contraceptives.
5. Chronic GT1b (2DAA arm) or Chronic GT 1 (1a or 1b) (3DAA arm) infection as documented by one or more measurements of serum HCV RNA greater than or equal to 2,000 IU/mL during screening and at least one of the following:

   1. A positive anti-HCV antibody, HCV RNA, or HCV genotype test result greater than or equal to 12 months prior to the baseline (Day 0) visit together with current positive HCV RNA or anti-HCV antibody test results.

Or

b. Positive HCV RNA test and anti-HCV antibody test results together with a liver biopsy consistent with chronic HCV infection or a liver biopsy performed before Day 0 with evidence of chronic hepatitis C infection disease, such as the presence of fibrosis.

6. HIV treatment status:

1. Documented HIV infection (defined by positive Western blot result or detectable HIV viral load), ARV untreated for >8 weeks preceding dosing and having either:

   1. A CD4 T-cell count greater than or equal to 500 cells/mm3 within 8 weeks of Day 0 or
   2. An HIV viral load less than 500 copies/mL with a stable CD4 count for at least 3 months
2. Documented HIV-1 (defined by positive western blot result or detectable HIV viral load) infection on a stable protocol-approved, ARV regimen for greater than or equal to 4 weeks prior to dosing and is expected to continue the current ARV regimen through the end of study with all of the following

   1. a CD4 T-cell count > 100 cells/mm3
   2. a documented plasma HIV-1 RNA level less than the level of detection measured at least twice in the 4 weeks preceding dosing. If the lower limit of detection of the local HIV-1 RNA result is >50 copies/mL (e.g., <70 copies/mL, the screening plasma HIV-1 RNA level cannot exceed 50 copies/mL).
   3. HIV ARV agents including only:

a. Raltegrativir plus one of the following

b. Tenofovir and emtricitabine or abacavir and lamivudine

7. Documentation of hepatitis C genotype 1b (2DAA arm) or GT 1 (1a or 1b) (3DAA arm) alone infection within 6 months prior to Day 0. HCV genotype/subtypes performed outside the NIH will be accepted for eligibility if performed using the Siemens LiPA v2.0 assay or an assay with equivalent performance in identifying the HCV genetype 1b (e.g., Abbott RealTime HCV Genotype II assay).

8. Liver biopsy obtained within 36 calendar months prior to the baseline (Day 0) visit to verify the presence or absence of cirrhosis, except as indicated below. If no recent (<36 months) liver biopsy is available, a liver biopsy may be performed prior to the baseline visit.

1. Cirrhosis is defined as any one of the following:

   1. Any biopsy showing cirrhosis (at any time, not restricted to the 36 calendar months prior to baseline visit).
   2. A FibroSUR[trademark] score, of >0.75 and an aspartate aminotransferase (AST) platelet ratio index (APRI) of >2 within the last year.
2. Absence of cirrhosis is defined as any one of the following:

   1. A liver biopsy performed within 36 calendar months of screening showing absence of cirrhosis.
   2. A FibroSUR[trademark] score, within the last year, of <0.48 and an APRI of <1.

      In the absence of a definitive diagnosis of presence or absence of cirrhosis by the criteria detailed above, a liver biopsy is required. The FibroSURE[trademark]test can be performed and the results can be used to determine the inclusion and exclusion criteria. Patients with Child Pugh B or C cirrhotics are excluded

   9. Ability to communicate effectively with the study investigator and other key personnel.

   10. Willingness to comply with the study restrictions and requirements.

   11. Opioid-dependent individuals must be participating in a supervised treatment program.

   12. Subjects must have an external primary care doctor (outside of the Clinical Center and the NIH) for their medical management.

   13. Willingness to have blood or tissue samples stored for future use to study liver disease and immune function.

   14. Willingness to undergo HLA typing.

   15. Otherwise healthy status as determined by medical history, physical examination, electrocardiogram (ECG), and clinical laboratory measurements performed at screening.

Contraception

The effects of ASV and DCV on the developing human fetus are unknown. For this reason, men and women of childbearing potential must agree to use adequate contraception as outlined in the inclusion and exclusion criteria prior to study entry and until 5 weeks (women ) and 14 weeks (men) after last dose of study medication. Hormonal contraception is NOT considered an effective form of birth control for female subjects on this study. Oral contraceptives are not as effective in women taking ASV and DCV so women cannot rely on this form of birth control to prevent pregnancy. Females of childbearing-age must have a negative pregnancy test result prior to receiving ASV and DCV. If a woman becomes pregnant or suspects of being pregnant during the course of the study, she should inform the study staff and her primary care physician immediately.

EXCLUSION CRITERIA

1. Current or prior history of any of the following:

   1. Clinically significant illness (other than HCV) or any other major medical disorder that may interfere with the subject treatment, assessment of compliance with the protocol; subjects currently under evaluation for a clinically-significant illness (other than HCV) are also excluded
   2. Gastrointestinal disorder with post-operative condition that could interfere with the absorption of the study drug
   3. Poor venous access interfering with required study blood collection
   4. Clinical hepatic decompensation (i.e.,-ascites, encephalopathy or variceal hemorrhage)
   5. Hepatic impairment (e.g., Child-Pugh class B [moderate] or Child-Pugh class C [severe])
   6. Solid organ transplantation
   7. Significant pulmonary disease, significant cardiac disease or porphyria.
   8. Unstable psychiatric disease (subjects with psychiatric illness that is well controlled on a stable treatment regimen or currently not requiring medication may be included)
   9. Any malignancy or its treatment that in the opinion of the PI may cause ongoing interference with host immunity; subjects under evaluation for malignancy are not eligible
   10. Significant drug allergy (such as anaphylaxis or hepatotoxicity)
   11. Chronic liver disease of a non-HCV etiology (e.g., hemochromatosis, Wilson s disease, alfa-1 antitrypsin deficiency, cholangitis)
2. Positive nucleotide sequence analyses of the NS5A gene for Y93H or L31M/V polymorphisms for the 2DAA arm only.
3. Positive test results at screening for hepatitis B virus (HBV) surface antigen (HBsAg) or HBV RNA (completed only if necessary to rule out chronic HBV)
4. Current use of non-protocol approved ARVs
5. A new AIDS-defining condition diagnosed within 30 days prior to date screening consent is signed or active serious infection (other than HIV and HCV), requiring parenteral antibiotics, antivirals or antifungals within 30 days prior to Day 0
6. Abnormal hematological and biochemical parameters at screening, unless the test has been repeated and at least one subsequent result is within the acceptable range prior to study drug administration, including:

   1. Neutrophil count <750 cells/mm3
   2. Hemoglobin level <9 g/dL
   3. Platelet count less than or equal to 50,000 cells/mm3
   4. Estimated glomerular filtration rate, calculated by the chronic kidney disease epidemiology collaboration formula: <50 mL/min/1.73 m^2
   5. ALT or AST level greater than or equal to10 times upper limit of normal (ULN)
   6. Serum lipase level greater than or equal to 1.5 times ULN at screening or during the screening period in a patient with symptoms of pancreatitis
   7. Total bilirubin level greater than or equal to 2.0 times ULN, except in subjects with Gilbert s syndrome
   8. Albumin level less than or equal to 3.0 g/dL
7. Donation or loss of blood of >400 mL within 8 weeks prior to the first dose of the study drugs
8. Poorly controlled diabetes as indicated by a screening glycosylated hemoglobin (HbA1c) >10
9. Known hypersensitivity to ASV, DCV or formulation excipients
10. Pregnant or breastfeeding
11. Screening or baseline with clinically significant ECG findings, or personal/first degree relative history of Torsade de pointes
12. Need for the use of the following medications from 21 days prior to the start of study drugs through the end of treatment:

    1. Hematologic stimulating agents, erythropoiesis stimulating agents (ESAs), granulocyte colony stimulating factor (GCSF), thrombopoeitin (TPO) mimetics
    2. Chronic systemic antineoplastic or immunomodulatory treatment including supraphysiologic doses of immunosuppressants such as corticosteroids (e.g., prednisone equivalent >10 mg/day for >2 weeks), azathioprine or monoclonal antibodies (e.g., infliximab)
    3. Investigational agents or devices for any indication
13. Previous treatment with an HCV protease inhibitor or any DAA
14. Medications for disease conditions excluded from the protocol (e.g.,- active cancer, transplantation) are not listed under the Concomitant medication section, and are disallowed from the study
15. Use of certain medications and herbal/natural supplements per PI discretion, expected to result in increases or decreases in exposure to study or non-study medications as listed in Section 5.5 while receving study medications and within five half-lives or 14 days [whichever is longer] of the first dose of study medications.
16. Co-enrollment Guidelines: Co-enrollment in other clinical trials is restricted, other than enrollment in observational studies or those evaluating the use of a licensed medication. Study staff should be notified of co-enrollment status, as it may require prior approval of the investigator

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-02; Primary Completion 2016-03 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Masur, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
NIH Biomedical Translational Research Information System

REFERENCES:
- [Background] Lok AS, Gardiner DF, Lawitz E, Martorell C, Everson GT, Ghalib R, Reindollar R, Rustgi V, McPhee F, Wind-Rotolo M, Persson A, Zhu K, Dimitrova DI, Eley T, Guo T, Grasela DM, Pasquinelli C. Preliminary study of two antiviral agents for hepatitis C genotype 1. N Engl J Med. 2012 Jan 19;366(3):216-24. doi: 10.1056/NEJMoa1104430. PMID 22256805
- [Background] Zeuzem S, Buti M, Ferenci P, Sperl J, Horsmans Y, Cianciara J, Ibranyi E, Weiland O, Noviello S, Brass C, Albrecht J. Efficacy of 24 weeks treatment with peginterferon alfa-2b plus ribavirin in patients with chronic hepatitis C infected with genotype 1 and low pretreatment viremia. J Hepatol. 2006 Jan;44(1):97-103. doi: 10.1016/j.jhep.2005.10.003. Epub 2005 Nov 7. PMID 16290907
- [Background] Kottilil S, Yan MY, Reitano KN, Zhang X, Lempicki R, Roby G, Daucher M, Yang J, Cortez KJ, Ghany M, Polis MA, Fauci AS. Human immunodeficiency virus and hepatitis C infections induce distinct immunologic imprints in peripheral mononuclear cells. Hepatology. 2009 Jul;50(1):34-45. doi: 10.1002/hep.23055. PMID 19551908

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HIV/HCV GT-1a/1b, 12 Wks ASV/DCV With BMS-791325 | HIV/HCV GT-1b, 24 Wks ASV/DCV
Started | 20 | 10
Completed | 20 | 9
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | HIV/HCV GT-1a/1b, 12 Wks ASV/DCV With BMS-791325 | HIV/HCV GT-1b, 24 Wks ASV/DCV | Total
Number analyzed (Participants) | 20 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 9 | 28
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 12 | 3 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 15 | 8 | 23
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 12 | 9 | 21
  White | 5 | 0 | 5
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Subjects Who Achieve Sustained Viral Response (SVR12) 12 Weeks After the Stop of Treatment Drugs
Description: The primary outcome was the percentage of patients with sustained viral response measured 12 weeks after the stop of treatment. The viral response was assessed by serum HCV RNA concentrations lower than 43 IU/mL - the lower limit of quantification.
Time Frame: 12 weeks after stop of treatment
Population: Subjects who received treatment drugs per arm as listed in the Outcome Measure Description
Measure: Number; unit: Percentage of subjects
Arm/Group | HIV/HCV GT-1a/1b, 12 Wks ASV/DCV With BMS-791325 | HIV/HCV GT-1b, 24 Wks ASV/DCV
Number analyzed (Participants) | 20 | 10
Percentage of subjects | 90 | 80

ADVERSE EVENTS:
Arm/Group | HIV/HCV GT-1a/1b, 12 Wks ASV/DCV With BMS-791325 | HIV/HCV GT-1b, 24 Wks ASV/DCV
Serious Adverse Events (participants affected / at risk) | 3/20 | 5/10
Other Adverse Events (participants affected / at risk) | 6/20 | 3/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HIV/HCV GT-1a/1b, 12 Wks ASV/DCV With BMS-791325 (N=20) | HIV/HCV GT-1b, 24 Wks ASV/DCV (N=10)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Paranoia (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HIV/HCV GT-1a/1b, 12 Wks ASV/DCV With BMS-791325 (N=20) | HIV/HCV GT-1b, 24 Wks ASV/DCV (N=10)
Fatigue (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Lipase increased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Panic disorder (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
One subject did not complete 24 weeks of study drug due to a HCV viral load rebound on treatment (at week 6) and was deemed a non-responder. This met the criteria for stopping study medications.

Nine subjects completed 24 weeks of therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes